CLINICAL TRIAL: NCT03528395
Title: Effectiveness of Commercial Video Games in Subacute Stroke Rehabilitation: Randomized Clinical Trial
Brief Title: Effectiveness of Commercial Video Games in Subacute Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital La Fuenfría (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP FUENFRÍA
Record Dates: First submitted 2018-05-05; First posted 2018-05-17 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: Balance; Baropodometry; Video games; Virtual reality
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomly distributed to a control group or experimental group using the QuickCalcs application of GraphPad Software.
  The following considerations will be taken into account:
  Control group: 8 weeks of conventional rehabilitation based on a task-oriented approach. Consisting of five weekly sessions of physical therapy and of occupational therapy, lasting 45 minutes each.
  Experimental group: 8 weeks of conventional rehabilitation provided identically as in the control group, plus virtual reality semi-immersive sessions. VR sessions will be applied following a protocol using commercial video games, three days a week (Monday, Wednesday and Friday) after the conventional rehabilitation sessions.
Who Masked: Investigator
Masking Description: All assessments will be made by blind evaluators with respect to the established study groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-immersive virtual reality (Experimental): 8 week protocol with semi-immersive virtual reality provided with the XBOX 360º video game console and its Kinect device. The commercial video games used will be: Kinect Sports I ®, Kinect Sport II ®, Kinect Joy Ride ® and Kinect Adventures ®.
  Interventions: Other: Semi-immersive virtual reality
- Conventional Rehabilitation (Active Comparator): Physical therapy and Occupational Therapy based on a task-oriented approach
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Semi-immersive virtual reality — Each participant will receive 24 additional sessions of semiinmersive virtual Reality therapy sessions on Monday, Wednesday and Friday, after realizing the conventional therapy sessions. The duration of each VR session will be gradually increased in time-intensity (5 minutes during the first week to 20 minutes during the last week) and motor requirements.
  Other Names: Commercial video games
  Arms: Semi-immersive virtual reality
Other: Conventional Rehabilitation — Conventional rehabilitation consisting of five weekly sessions of Physical therapy and Occupational Therapy, based on a task-oriented approach, lasting 45 minutes each.
  Other Names: Physical therapy and Occupational Therapy
  Arms: Conventional Rehabilitation

SUMMARY:
Stroke creats dependancy of patients due to various associated impairments. The use of low-cost technologies for neurological rehabilitation may be beneficial for the treatment of these patients.

DETAILED DESCRIPTION:
To determine the effectiveness of a structured protocol using semi-immersive virtual reality with commercial videogames for balance, postural control, functional independence, quality of life and motivation in patients who have suffered an ischemic and / or hemorrhagic stroke in subacute phase and are being treated in a mid-stay hospital.

Patients and methods: Randomized Controlled Trial. Simple blind. Control group will receive conventional therapy (physical therapy and occupational therapy) intervention being based on a task-oriented approach, with five weekly sessions of Physical Therapy and Occupational Therapy with duration of 45 minutes per session.

The experimental group will receive in addition to the above an experimental intervention during 8 weeks providing additional treatment using virtual reality semi-immersive complement is added by means of commercial video games implemented with the Xbox 360º video game console in conjunction with the Kinect device.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CVA in subacute ischemic or hemorrhagic type.
* NIHSS scale score less than 20.
* MoCA test with scores equal to or greater than 14 (mild cognitive impairment or absence of cognitive impairment).
* Modified Rankin scale between 0-4.
* Patients with the ability to maintain autonomous sitting and standing with or without aids.
* Patients who have received the information document of the study and signed the informed consent form.

Exclusion Criteria:

* NIHSS scale scores greater than 21 .
* MoCA test with score lower than 14.
* Modified Rankin scale between 5-6.
* Patients without the ability to maintain autonomous sitting.
* Patients who refused to sign the informed consent form.
* Hospital discharge expected at the beginning of the study.
* Patients who at any time have shown worsening of the general state, disinterest or desire to leave the study.

  * Pathologies susceptible to worsening or contraindication with virtual reality devices and commercial video games:

    * Photosensitive epilepsy.
    * Modified Ashworth scale greater than 2.
    * Moderate-severe cognitive impairment.
    * Visual alterations.
    * Non-collaborating patient.
    * Behavioral alterations.
    * Refusal to treatment with VR systems.
    * Presence of other neurological pathologies.
    * Other cardiovascular diseases that contraindicate physical exercise.
  * Visual or auditory, musculoskeletal, bone or joint alterations in acute or chronic phase that could influence the primary pathology.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Timed get up and go | eight weeks
  It is a test used to evaluate functional mobility and balance, adapted and translated into Spanish. The patient must get up from a chair, walk three meters in a straight line, turn and return to sit in the chair. The valuation is quantified from 1 to 5: 1- normal, and 5- fall hazard during the test. At present study was conducted supervised by two people that were placed laterally to the patient.

SECONDARY OUTCOMES:
Tinetti scale | eight weeks
  Scale validated in the context of stroke and whose score maximum for balance is 16 points, and 12 for gait. The higher the score, the lower risk of falls (less than 19 points on the scale total implies a high risk of falls; the risk is moderate with scores of 19 to 24).
Baropodometry | eight weeks
  The T-plate ® pedometer provides information on the pressure exerted by each point of the sole of the foot, distribution and plantar symmetry through a static test in the standing position. This test registers the center of pressures at a given moment, offering information on the distribution load (%) and the support surface.
Static Posturography | eight weeks
  Postural and static balance in standing was assessed through lateral and anteroposterior movement of the center of pressures in the x and y axes, in centimeters and square centimeters. Tests carried out were the Romberg test with open eyes, in which the patient remains on the platform and try to maintain balance during 30 seconds, and the Romberg test with eyes closed, in which the patient remains on the platform with closed eyes and tries to keep their balance for 30 seconds.
Functional reach test | eight weeks
  This test was used to detect alterations of the postural control and balance. The patient is placed standing holding the arm with the shoulder at 90 ° flexion, with a clenched fist, then realizes a maximum anterior reach without moving the feet of the ground. The maximum forwards distance without any supports is measured. A rigid tape measure with a leveler was used of a rule and bubble level calibrated bubble adhered to a mirror located on the wall. Patients able to perform this test were located with the healthy side next to the mirror, without direct contact. The result is registered in centimeters, measuring the distance between the initial and final position.
Modified Rankin scale | eight weeks
  Assesses the degree of physical disability after a stroke assigning a subjective score from 1 to 5. It is a very useful tool, validated and translated, to categorize functional level. It was used as a valuation tool pre and post intervention to describe changes in the level of functional independence of the patient after the experimental intervention.
Barthel index | eight weeks
  In order to assess functional independence, the Barthel index, indicated to evaluate the activities of daily life and validated in the Stroke context, translated and adapted to Spanish. It consists of 10 items with a range of score between 0 and 100 (with lower score, greater dependency).
EQ-5D Questionnaire | eight weeks
  The quality of life related to health was evaluated through the EuroQoL 5D. It is a test self-administered, generic, adapted to Spanish, in which health status is assessed in five dimensions (mobility, personal care, activities daily, pain / discomfort and anxiety / depression), and includes an optimal visual analog scale to assess the state of health at the time of registration (0-100).
Cano-Mañas scale | eight weeks
  The level of motivation, self-esteem and adherence to intervention was assessed using the Cano- Mañas. It is a Likert scale prepared by the research team and made since there is no validated instrument and translated that met the specific needs required. The first week of intervention was administered experimental and at the end of the eight weeks. It included 16 items (five motivation items, five of self-esteem and six of adhesion to the intervention). The scores were measured between 1 and 6: 1- very much in agreement; 5- strongly disagree; and 6-I have no opinion.

CONTACTS AND LOCATIONS:
Overall Officials: MªJosé Cano Mañas, PhD program, Principal Investigator — Hospital La Fuenfría; Roberto Cano de la Cuerda, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Hospital La Fuenfría, Cercedilla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cano-Manas MJ, Collado-Vazquez S, Cano-de-la-Cuerda R. [Commercial video games in the rehabilitation of patients with sub-acute stroke: a pilot study]. Rev Neurol. 2017 Oct 16;65(8):337-347. Spanish. PMID 28990643
- [Derived] Cano-Manas MJ, Collado-Vazquez S, Rodriguez Hernandez J, Munoz Villena AJ, Cano-de-la-Cuerda R. Effects of Video-Game Based Therapy on Balance, Postural Control, Functionality, and Quality of Life of Patients with Subacute Stroke: A Randomized Controlled Trial. J Healthc Eng. 2020 Feb 13;2020:5480315. doi: 10.1155/2020/5480315. eCollection 2020. PMID 32148744